CLINICAL TRIAL: NCT00448617
Title: Cigarette Smoke and Susceptibility to Influenza Infection
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Hamner Institutes for Health Sciences (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Terry Noah, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Other Study IDs: 05-PED-1094
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: live attenuated influenza virus; inflammation; flu vaccine; FluMist; smokers
MeSH Terms: conditions — Inflammation; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal lavage fluid, urine, blood, nasal epithelial tissue from subjects who consent to have excess samples stored in our repository
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be a descriptive comparison of the effects of live attenuated influenza virus (FluMist) on nasal inflammation and oxidative stress in healthy young adults who are not exposed to smoke vs smokers. It is hypothesized that passive exposure to second-hand smoke (SHS) results in increased susceptibility to the effects of influenza virus in nasal epithelium in humans and that these effects are mediated by SHS-induced oxidative stress

DETAILED DESCRIPTION:
Epidemiologic evidence supports a significant relationship between passive cigarette smoke exposure and increased risk for viral respiratory illnesses. Published and preliminary data suggest that airborne pollutants including tobacco smoke increase susceptibility of respiratory epithelium to infection with influenza A and that this effect is at least partially mediated by oxidative stress. However, no studies have specifically looked at the interaction between smoking and the effects of influenza virus in human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* healthy nonsmoking who are rarely exposed to SHS OR smokers

Exclusion Criteria:

* pregnancy or nursing;
* history of egg allergy;
* aspirin therapy;
* asthma;
* immunodeficiency (HIV or other);
* on immunosuppressive drugs including corticosteroids;
* history of Guillain-Barre Syndrome;
* any chronic medical condition;
* febrile and/or respiratory illness within past 3 weeks prior to entry into study;
* prospective subjects with high baseline antibody titers against influenza will be excluded because they may be less likely to develop viral replication with LAIV.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. smokers
  2. nonsmokers who are NOT exposed to SHS
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2006-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Nasal responses of healthy adult volunteers not routinely exposed to SHS vs responses of smokers, to live attenuated influenza virus. | 5-8-weeks

SECONDARY OUTCOMES:
Compare replication of live attenuated influenza virus (LAIV) in nasal epithelium of seronegative healthy adult volunteers not routinely exposed to SHS vs. smokers. | 5-8 weeks
In the setting of LAIV infection, compare markers of oxidant stress and mucosal inflammation in nasal epithelium of healthy adult volunteers not routinely exposed to SHS vs. smokers | 5-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Center for Environmental Medicine, Asthma and Lung Biology — http://www.med.unc.edu/cemalb/